CLINICAL TRIAL: NCT03947879
Title: The Effect of Pharmaceutical Grade L-glutamine (Endari) on Glycemic Control in Patients With Diabetes Mellitus Type II
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hawaii Pacific Health (Other)
Responsible Party: Principal Investigator, Charles R Zerez, PhD, MD, Internal Medicine Physician, Hawaii Pacific Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-119
Record Dates: First submitted 2019-04-17; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- L-glutamine (Experimental): Treatment with L-glutamine for 3 months.
  Interventions: Drug: L-glutamine
- No L-glutamine (Experimental): No L-glutamine for 3 months.
  Interventions: Other: No L-glutamine

INTERVENTIONS:
Drug: L-glutamine — 15 g of L-glutamine twice daily by mouth for 3 months.
  Other Names: Endari
  Arms: L-glutamine
Other: No L-glutamine — The same patients will be given no L-glutamine for 3 months.
  Arms: No L-glutamine

SUMMARY:
The study is an initial non-blinded, non-placebo controlled trial to determine the efficacy of L-glutamine in lowering blood sugar in patients with diabetes mellitus type II without sickle cell anemia.

DETAILED DESCRIPTION:
The protocol will consist of starting patients on 15 g of L glutamine twice daily by mouth. This is the same dose that is used to treat patient with sickle cell anemia. They will be given this medication for a total of 3 months. Their other medications will remain the same. At the conclusion of the 3 months, the patients will be taken off of the glutamine and will continue their other medications. The investigators will monitor the patients an additional 3 months (6 months after the initiation of the study) off the L-glutamine. In this manner, the investigators will have a washout period. The outcome will be a comparison of the results before the initiation of the L-glutamine, to the results after treatment, and after the washout.

Data analysis will consist of comparing the patient's fasting glucose and hemoglobin A1c values. The investigators will also check the levels of fructosamine. This is a standard test that is done in any clinical laboratory. To help determine the mechanism for the L-glutamine effect, the investigators will also measure the complete blood count, chemistry panel, hepatic function panel, urine micro-albumin, patients' weight, and waist circumference. The investigators will use the Student t-test for statistical analysis. Significance will be tested at the 0.05 level.

The investigators will collect demographic information on the patients in the study. Age, sex, duration of diabetes, smoking history, and race will be noted. The investigators will use regression analysis to determine whether these factors have any effects on the observed results.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of diabetes mellitus type II
* Patient of Straub Medical Center, Internal Medicine Clinic

Exclusion Criteria:

* Renal and liver impairment ( GFR less than 40)
* Transaminitis (elevation of AST of ALT more than 2 fold)
* Patient with sickle cell anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in fasting glucose | 3 months and 6 months
  Change in fasting glucose
Change in hemoglobin A1c | 3 months and 6 months
  Change in hemoglobin A1c

SECONDARY OUTCOMES:
Change in fructosamine | 3 months and 6 months
  Change in fructosamine level
Change in complete blood count | 3 months and 6 months
  Change in complete blood count
Change in blood chemistry | 3 months and 6 months
  Change in blood chemistry
Change in hepatic function | 3 months and 6 months
  Chang e in hepatic function
Change in microablbumin | 3 months and 6 months
  Change in urine microalbumin
Change in weight | 3 months and 6 months
  Change in weight
Change in waist circumference | 3 months and 6 months
  Change in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Charles Zerez, MD, PhD, Principal Investigator — Straub Medical Center

IPD SHARING:
Plan to Share IPD: No